CLINICAL TRIAL: NCT06685042
Title: Anti-CD19 CAR T-Cell Therapy in Refractory Systemic Autoimmune Diseases
Acronym: CATARSIS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, D'Agostino Maria Antonietta, Full Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6192; 2024-511293-74-01 (EU CTIS Number)
Record Dates: First submitted 2024-10-25; First posted 2024-11-12 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Lupus Erythematosus, Systemic; System; Sclerosis; ANCA Associated Vasculitis; Dermatomyositis; Polymyositis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Diffuse; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Dermatomyositis; Polymyositis | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-CD19 CAR T cell (Experimental): Single intravenous infusion of 1 x 106 /kg body weight CAR T cell ("CD19-CAR_Lenti" )
  Interventions: Biological: CAR T cell

INTERVENTIONS:
Biological: CAR T cell — The investigational medicinal product (IMP) "CD19-CAR_Lenti" consists of autologous CD19 Chimeric Antigen Receptor (CAR) transduced CD4/CD8 enriched T cells, derived from a leukapheresis product and processed by using the CliniMACS Prodigy® device (Miltenyi Biotec). CD19-CAR_Lenti is a suspension of fresh CD4/CD8-enriched CD3+ T cells that have been genemodified with a self-inactivating (SIN) lentiviral vector expressing a CAR directed against human CD19. The SIN lentiviral vector is derived from clinically validated viral vectors described in the literature with a fully characterized sequence.

SUMMARY:
The CATARSIS study explores the use of anti-CD19 CAR T-cell therapy as a novel approach for treating refractory systemic autoimmune diseases, specifically SLE, SSc, DM/PM, and AAV. These life-threatening conditions often resist current therapies, and B cells play a key role in their pathogenesis. The study employs CD19-CAR_Lenti, an autologous CAR T-cell product targeting CD19-positive B cells, aiming to reduce inflammation and autoimmunity. This open-label, single-dose, phase I basket trial will assess the safety, feasibility, and preliminary efficacy of CAR T-cell therapy, focusing on adverse events, infection rates, and overall response at 24 weeks. Eight participants will be included.

DETAILED DESCRIPTION:
In recent years, B cells have become more appreciated as major players and also as therapeutic targets in systemic autoimmune diseases. Systemic autoimmune diseases, such as Systemic Lupus Erythematosus (SLE), Systemic Sclerosis (SSc), Dermatomyositis/Polymyositis (DM/PM), and ANCA Associated Vasculitis (AAV) are among the most life-threatening diseases. Even though clinical presentation and organ involvement may be different, these diseases share common pathways of B cell activation. Despite the substantial advances in their management, some patients with systemic autoimmune diseases fail to respond to the current state-of-the art therapies, and are at high risk for severe organ failure and even death. Therefore, new treatments for such refractory cases are urgently needed.

A strong preclinical rationale supports the use of anti-CD19 CAR T cells in systemic autoimmune disease. Experimental animal models back the concept that anti-CD19 CAR T cell therapy could be a powerful approach to target autoimmunity and inflammation in B cell mediated autoimmune disease. "CD19-CAR_Lenti" (the ATMP) consists of autologous CD19 Chimeric Antigen Receptor (CAR) transduced CD4/CD8 enriched T cells, derived from a leukapheresis product and processed at Officina Farmaceutica of IRCCS Ospedale Pediatrico Bambino Gesù through a validated process by using the CliniMACS Prodigy® device. CD19-CAR_Lenti is a suspension of fresh CD4/CD8- enriched CD3+ T cells that have been gene-modified with a self-inactivating (SIN) lentiviral vector expressing a CAR directed against human CD19.

CATARSIS is a basket study on four prototypic systemic autoimmune diseases, which a) show a severe life-threatening disease course, b) are associated with a current high unmet need for treatment, c) show an involvement of B lymphocytes in disease pathogenesis and d) respond at least partially to treatment with B cell depleting antibodies.

The investigators will conduct a prospective, open-label, single-dose, non-randomized, interventional phase I clinical study, using a "basket" design, to assess the safety, feasibility, and preliminary efficacy of ex vivo generated autologous anti-CD19 CAR T cells targeting a common pathogenic pathway (activated B cells and plasmablasts) in subjects with severe, treatment-failure systemic autoimmune disease (SLE, SSc, DM/PM and AAV).

In particular, the investigators will assess incidence and grading of severity of Cytokine Release Syndrome (CRS) and of CAR T cell Associated Neurotoxicity Syndrome (ICANS) within the first 4 weeks after ATMP administration, incidence and severity of infections and leukopenia and/or hypogammaglobulinemia during the entire study period (24 weeks), and overall Response Rate (ORR) at week 24 based on specific disease activity composite indexes, each of them validated for the specific disease.

Duration of B cell depletion in the peripheral blood, duration of persistence of CAR T cells in the peripheral blood, and changes in the levels of disease-associated serum autoantibodies will be assessed as well through specific laboratory measurements.

A total of 8 subjects with B cell-mediated autoimmune disease will be included in the CATARSIS study, following a Bryant and Day two stages design. Subjects will receive a single intravenous infusion of 1 x 10^6 /kg body weight CAR T cell. Recruitment and outpatient visits will be performed in the UOC Reumatologia - Dipartimento di scienze dell'Invecchiamento, Ortopediche e Reumatologiche (FPG) and Dipartimento Oncoematologia, Terapia Cellulare, Terapie Geniche e Trapianto Emopoietico (OPBG). Treatment and pre-treatment specific procedures (leukapheresis, lymphodepletion) of subjects and the inpatient visits will be performed in the UOC Ematologia e Trapianto di cellule staminali emopoietiche - Dipartimento di diagnostica per Immagini, Radioterapia Oncologica ed Ematologia (FPG) and Dipartimento Oncoematologia, Terapia Cellulare, Terapie Geniche e Trapianto Emopoietico (OPBG) by trained investigators. ATMP manufacturing will be performed in a certified facility at Officina Farmaceutica, IRCCS Ospedale Pediatrico Bambino Gesù, under licenses by local regulatory authorities and highest technical standards.

ELIGIBILITY:
Inclusion criteria

* General

  1. Subjects must understand and voluntarily sign an informed consent form, including written consent for data protection;
  2. Adults aged ≥ 18 years and < 65 years at time of consent;
  3. Male subjects, unless surgically sterile, must agree to use two acceptable methods for contraception (e.g., spermicide and condom) during the trial and refrain from fathering a child starting from the time of signing the Informed Consent Form (ICF) until 12 months after dosing of the IMP;
  4. Females of childbearing potential (FCBP) must have a negative urine pregnancy test at screening and must agree to use a highly effective contraceptive method (Pearl index <1) starting from the time of signing the ICF and for 12 months after dosing of the IMP;
  5. Must be able to adhere to the study visit schedule and other protocol requirements;
  6. Double vaccination (2 doses) against SARS-CoV-2 or SARS-CoV-2 within the last 6 months.
* SLE subjects

  a) Fulfilling the 2019 ACR/EULAR classification criteria of SLE; b) Presence of anti-dsDNA, anti-histone, anti-nucleosome or anti-Sm antibodies; c) Active disease at screening, defined as ≥1 organ system with a British Isles Lupus Assessment (BILAG) A score (severe disease activity) or ≥2 organ systems with a BILAG B score (moderate disease activity); d) Insufficient response to glucocorticoids and at least 2 of the following treatments: hydroxychloroquine, mycophenolate mofetil, belimumab, methotrexate, rituximab.
* SSc subjects

  1. Fulfilling the 2013 ACR/EULAR classification criteria of SSc;
  2. Diffuse SSc with respective autoantibody profile;
  3. Signs for fast progression including i) disease duration ≤5 years (from onset of first non-Raynaud manifestation), ii) mRSS score 10-35 at screening, iii) elevated acute phase reactant levels (CRP ≥ 6 mg/L, ESR ≥ 28mm/h or platelet count ≥ 330 000/mm3), iii) mRSS increase ≥ 3 units or involvement of one new body area or mRSS increase ≥ 2 units in one body area or ≥1 tendon friction rub over 6 months;
  4. Insufficient response to glucocorticoids and to at least 2 of the following treatments:

mycophenolate mofetil, azathioprine, nintedanib, methotrexate, rituximab.

* DM/PM subjects

  a) Fulfilling the 2017 ACR/EULAR classification criteria for probable or definite DM or PM57, b) Muscle weakness as defined by MMT < 142 and 2 of the following criteria: VAS patients Global ≥ 2 cm, VAS physician Global ≥ 2 cm, HAQ > 0.25, at least one muscle enzyme >1.3 times upper limit of normal, VAS global extra muscular activity ≥ 2 cm; c) Presence of at least one myositis-specific antibody; d) Insufficient response to glucocorticoids and to at least 2 of the following treatments: mycophenolate mofetil, ciclosporin A, tacrolimus, methotrexate, rituximab, and intravenous immunoglobulins.
* AAV subjects

  1. Fulfilling the 2022 ACR/EULAR classification criteria for MPA/GPA/EGPA,
  2. Presence of ANCA to either proteinase 3 or myeloperoxidase;
  3. At least one major or three non-major items or at least two renal items of hematuria and proteinuria on the BVAS;
  4. Failure of at least 1 of the following treatments: glucocorticoids, cyclophosphamide, or B-cell targeting therapy.

Exclusion criteria

* Clinically suitability for a less burdensome and/or approved therapeutic approach, as judged by the investigator;
* ANC < 1.000/mm3, ALC < 500/mm3 or hemoglobin < 8 g/dl, absolute CD3+ T cell count ≤100/µl;
* Evidence of significant and uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results.
* Relevant cardiovascular disease: recent history of myocardial infarction, cardiac angioplasty or stenting, unstable angina, significant arrhythmia, congestive heart failure, or left ventricular ejection fraction < 50%, as determined by echocardiography
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study;
* Impaired renal function, i.e., eGFR < 30 ml/min;
* Patients with evidence on thorax CT of advanced fibrotic interstitial lung disease and whose latest pulmonary function test showed a Forced Vital Capacity (FVC) < 40% of predicted or a Diffusing Capacity for Carbon Monoxide (DLCO) < 30% of predicted
* Any concomitant severe active infection, including HIV (even with negative viral load), active hepatitis B (either positive for Hepatitis B core antibody [HBcAb] or positive hepatitis B surface antigen [HBsAg] and NAT tests) and/or C (<12 weeks between achievement of a sustained virological response to the specific treatment and apheresis) according to the American Association for the Study of Liver Diseases guidelines, SARS-CoV 2 (COVID 19), or active tuberculosis as defined by a positive Quantiferon TB-test. If the presence of latent tuberculosis is established, then treatment according to local guidelines must have been initiated before enrolment;
* Pregnant or lactating females;
* Known hypersensitivity to either any drug components or any auxiliary medicinal products scheduled during trial participation, including during lymphodepletion;
* Malignancy in the last 5 years before screening. The inclusion of patients with previously completely resected carcinoma in situ who have not required treatment other than surgery is allowed.
* Previous CAR T cell administration;
* A therapeutic schedule not compatible with the wash-out requirements for the leukapheresis procedure (section 5.8.1 of CSP) and the medications permitted during the study (section 7.11 of CSP);
* Concurrent treatment with other investigational agents or participation in other investigational trials.
* Treatment, as part of an investigational clinical trial, with an experimental product with a definite or potential effect on T or B-cells in the previous 2 years.
* Requirement for immunization with live vaccine during the study period or within 14 days preceding leukapheresis;
* Subjects who are younger than 18 years or are incapable of understanding the aim, importance, and consequences of the study and giving legal informed consent;
* Have a history of alcohol or substance abuse within the preceding 6 months that, in the opinion of the Investigator, may increase the risks associated with study participation or study agent administration or may interfere with the interpretation of results;
* Subjects who possibly are dependent on the Sponsor, the Principal Investigator, or the Investigator (e.g., family members).
* Limited to patients diagnosed with SLE: patients with a history of severe central nervous system (CNS) involvement, including those who have presented aseptic meningitis, cerebral vasculitis, cerebrovascular disease, demyelinating syndrome, myelopathy, seizure disorder, status epilepticus, and severe lupus headache, will be excluded.
* Patients meeting the classification criteria for multiple connective diseases such as overlapping SLE and Sjogren's Syndrome (SS) or SLE and Rheumatoid Arthritis (RA) and patients diagnosed with Mixed Connective Tissue Disease (MCTD).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects experiencing a CRS or an ICANS | 4 weeks
  The first safety outcome variable will be measured as the number of subjects experiencing a Cytokine Release Syndrome (CRS) or an (Immune Effector Cell-associated Neurotoxicity Syndrome) ICANS within the first 4 weeks after ATMP administration in relation to the number of subjects enrolled in the study.
Incidence of infections, leukopenia and/or hypogammaglobulinemia | 24 weeks
  The second safety outcome variable will be measured as the incidence of infections, leukopenia, and/or hypogammaglobulinemia during the entire study period in relation to the number of subjects enrolled in the study.
Overall Response Rate | 24 weeks
  The efficacy outcome variable, Overall Response Rate (ORR), is defined as the ratio between the number of subjects experiencing a response at week 24 and the total number of enrolled subjects.
  A response to treatment will be considered at week 24 as:
  * SLE: Fulfillment of DORIS remission criteria of SLE.
  * SSc: No progression of interstitial lung disease with worsening of FVC (>10%) or worsening of FVC (5-10%) plus an increase in respiratory symptoms or worsening of FVC (5-10%) plus progression of high-resolution computed tomography changes after 24 weeks.
  * DM/PM: 2016 ACR/EULAR Moderate or Major Response.
  * AAV: Birmingham vasculitis activity score (BVAS) of 0.

SECONDARY OUTCOMES:
Time of persistence of CAR T cells | 24 weeks
  Time of persistence of CAR T cells in the peripheral blood is defined as the time elapsed from the date of the study intervention and the date of disappearance of CAR T cells. CAR T cells will be identified as proportion of CAR+ cells relative to total CD3+ cells (0-100%) and in absolute number (cells per milliliter of peripheral blood).
Time of absence of B cells in the peripheral blood | 24 weeks
  Time of absence of B cells in the peripheral blood is defined as the time elapsed from the date of the study intervention and the date of the rise of B cells after the intervention-induced nadir. B cells will be identified as proportion of CD19+ cells relative to total lymphocytes (0-100%) and in absolute number (cells per milliliter of peripheral blood).
Time to the disappearance of autoantibodies in the serum | 24 weeks
  Time to the disappearance of autoantibodies in the serum is defined as the time elapsed from the date of the study intervention and the date of negativization of disease-specific autoantibodies. The negativity of an autoantibody is defined as its detection at a concentration (AU/mL) below the lower limit of positivity, according to the laboratory's reference ranges.

OTHER OUTCOMES:
B cell receptor and T cell receptor repertoire | 24 weeks
  B cell receptor and T cell receptor usage as determined by sequencing analysis of circulating B cells and T cells in the peripheral blood at screening and week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Antonietta D'Agostino, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Lazio, Italy